CLINICAL TRIAL: NCT01600235
Title: Safety and Efficacy of Therapeutic Induced Hypertension in Patients With Acute Non-cardioembolic Ischemic Stroke: A Multicenter, Randomized, Open Label, Prospective, Phase 3 Study
Brief Title: Safety and Efficacy of Therapeutic INduced HYPERTENSION in Acute Non-cardioembolic Ischemic Stroke (SETIN-HYPERTENSION)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Inje University (Other); Gyeongsang National University Hospital (Other); Seoul National University Bundang Hospital (Other); Keimyung University Dongsan Medical Center (Other); Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Oh Young Bang, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-01-023
Record Dates: First submitted 2012-05-13; First posted 2012-05-17 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Stroke, Acute; Progressing Stroke
Keywords: Stroke, ischemic; Progression; Induced-hypertension; Phenylephrine
MeSH Terms: conditions — Stroke; Ischemic Stroke; Disease Progression | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenylephrine (Experimental): Phenylephrine induced-hypertension arm
  Interventions: Drug: Phenylephrine
- Conventional treatment (No Intervention): Control arm

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine (0.12mg/mL) Starting dose: 10cc/hr Titration: increase 10cc/hr every 30-60min, maximum 160cc/hr rate: increase systolic blood pressure (SBP) 10-25mmHg /hr Target: initially 20% increase of initial SBP, up to improving NIHSS score or SBP 200mmHg
  Arms: Phenylephrine

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the induced hypertension using phenylephrine in patients with noncardioembolic ischemic stroke.

The investigators hypothesized that phenylephrine induced-hypertension can result in good clinical response without serious complications in patients with noncardioembolic ischemic stroke.

DETAILED DESCRIPTION:
See below

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke confirmed by diffusion-weighted imaging (DWI) performed within 24 hours of symptom onset or symptom worsening(defined by a 2-point or more increase in NIH stroke scale (NIHSS)score including one or more increase in the motor score of affected upper and lower limbs in NIHSS during hospitalization or clear history of symptom worsening judged by investigator before hospitalization) confirmed by DWI performed within 24 hours of aggravation.
* Baseline NIHSS score 4-18 points
* Alert mental status
* Newly developed paresis, aphasia, or neglect

Exclusion Criteria:

* Patients underwent recanalization therapy
* Systolic blood pressure >170 mmHg at baseline
* Patients with history or at risk of hemorrhagic stroke
* History of significant arrhythmia (e.g. atrial fibrillation)
* Unable to perform MRI scans or undergo MRI scans > 24 hours of symptom onset or progression
* Large cortical infarction on DWI (more than 1/2 of middle cerebral artery territory)
* 3 or more cortical microbleeds on gradient-echo MRI
* Coronary artery disease, congestive heart failure, or hypertrophic cardiomyopathy
* Anticoagulation therapy (phenylephrine group only)
* Patients with high-risk cardioembolic sources
* Cervical or cerebral artery dissection or unruptured aortic/cerebral arterial aneurysm
* Decreased consciousness
* Pregnant or Lactating patient
* Seizure at stroke onset
* Life expectancy < 6 months
* Pre-stroke modified Rankin scale (mRS) >= 2
* Patients without informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Day 0 and Day 7
  2 points improvement in NIH stroke scale (NIHSS) between days 0 and 7

SECONDARY OUTCOMES:
Secondary efficacy outcome | Day 90 for 1, 2 and Day 7 for 3
  1. modified Rankin scale (mRS)≤ 2 at day 90
  2. modified Bathel index (mBI)≥ 90 at day 90
  3. Infarct growth or new ischemic lesion on follow-up MRI
Major safety outcome | From date of randomization until the date of first documented progression by intracranial hemorrhage or cerebral edema, date of myocardial infarction, or date of death from any cause, whichever came first, assessed up to 3 months
  1. Symptom aggravation by intracranial hemorrhage or cerebral edema (Clinical deterioration causing an increase in the NIHSS score of more than or equal to 4 points and if the hemorrhage or edema was liley to be the cause of the clinical deterioration)
  2. Myocardial infarction
  3. death from any cause
Minor safety outcome | From date of randomization until the date of first documented intracranial hemorrhage on follow-up MRI, or date of first documented side effects, whichever came first, assessed up to 3 months
  1. Intracranial hemorrhage on follow-up MRI
  2. Side effects including headache, arrhythmia, chest pain, dysuria, or gastrointestinal hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Bang OY, Chung JW, Kim SK, Kim SJ, Lee MJ, Hwang J, Seo WK, Ha YS, Sung SM, Kim EG, Sohn SI, Han MK. Therapeutic-induced hypertension in patients with noncardioembolic acute stroke. Neurology. 2019 Nov 19;93(21):e1955-e1963. doi: 10.1212/WNL.0000000000008520. Epub 2019 Oct 23. PMID 31645472